CLINICAL TRIAL: NCT02000531
Title: Ensure Extension Study to Assess the PFS of First-Line Erlotinib (Tarceva®) and Erlotinib After the Time of Disease Progression in Chinese Population Enrolled in the Ensure Trial
Brief Title: Progression Free Survival (PFS) Using Erlotinib for Non-Small-Cell Lung Cancer (NSCLC) in Chinese Population
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML29028
Record Dates: First submitted 2013-11-27; First posted 2013-12-04 (Estimated); Results first posted 2016-01-13 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2015-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non-small-cell lung cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Drug Therapy; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Erlotinib-Chemotherapy (Experimental): Erlotinib in first-line treatment, followed by chemotherapy in the second-line treatment
  Interventions: Drug: Erlotinib; Drug: Chemotherapy
- Chemotherapy-Erlotinib (Active Comparator): Chemotherapy in first-line treatment, followed by erlotinib in the second-line treatment
  Interventions: Drug: Erlotinib; Drug: Chemotherapy

INTERVENTIONS:
Drug: Erlotinib — 150 mg oral dose of erlotinib given once daily
  Other Names: Tarceva
Drug: Chemotherapy — Cisplatin (75 mg/m^2 intravenously [IV]) on Day 1 and gemcitabine (1250 mg/m^2 IV) on Days 1 and 8 of 3-week chemotherapy cycles until disease progression, unacceptable toxicity or up to 4 cycles (whichever comes first)
  Other Names: Gemcitabine/Cisplatin

SUMMARY:
This trial is an extension to ENSURE, a study of erlotinib versus gemcitabine/cisplatin combination chemotherapy as the first-line treatment for patients with non-small-cell lung cancer (NSCLC) with mutations in the tyrosine kinase domain of EGFR.

This study is designed to examine the efficacy of erlotinib versus gemcitabine/cisplatin as a second-line treatment in NSCLC patients from the ENSURE trial (NCT01342965). Patients previously treated with gemcitabine/cisplatin will be given erlotinib daily until disease progression or unacceptable toxicity occurs. Patients previously treated with erlotinib will be given cisplatin on Day 1 and gemcitabine on Days 1 and 8 of 3-week chemotherapy cycles until disease progression, unacceptable toxicity or up to 4 cycles (whichever comes first).

ELIGIBILITY:
Inclusion Criteria:

* Participant in ENSURE trial
* Disease progression during first-line treatment

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- China (9):
  - Beijing
  - Changchun
  - Chongqing
  - Fuzhou
  - Guangzhou
  - Nanjing
  - Shanghai
  - Shantou
  - Wuhan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erlotinib-Chemotherapy | Chemotherapy-Erlotinib
Started | 21 | 24
Safety Population | 21 | 24
Completed | 17 | 16
Not Completed | 4 | 8
Not completed — Lost to Follow-up | 1 | 0
Not completed — Discontinued due to data cut-off | 3 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Erlotinib-Chemotherapy | Chemotherapy-Erlotinib | Total
Number analyzed (Participants) | 21 | 24 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 18 | 35
  >=65 years | 4 | 6 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (8.20) | 57.0 (11.32) | 57.3 (9.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 9 | 14 | 23
Region of Enrollment [Number; unit: participants]
  China | 21 | 24 | 45

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Based on Well-documented and Verifiable Progression Events
Description: Progression free survival is defined as the time of randomization in ENSURE study to progressive disease (PD) while on second-line treatment or death from any cause, whichever occurred first during the second-line treatment.
Time Frame: within 3 years, 9 months (data cut-off December 2014)
Population: Intention to treat population, defined as all participants enrolled in this extension study
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Erlotinib-Chemotherapy | Chemotherapy-Erlotinib
Number analyzed (Participants) | 21 | 24
Months | 26.3 [19.8 to 34.0] | 23.4 [17.8 to 39.0]
Statistical Analysis 1: Comparison: Erlotinib-Chemotherapy vs Chemotherapy-Erlotinib; Test type: Superiority or Other; p > 0.05, Log Rank; Hazard Ratio (HR) = 1.26, 95% CI 2-sided [0.61 to 2.62]

2. Secondary Outcome: Participants With Adverse Events
Time Frame: start of second-line treatment to data cut-off in December 2014 (within 12 months)
Population: Safety Population, defined as all participants enrolled in this extension study
Measure: Number; unit: participants
Arm/Group | Erlotinib-Chemotherapy | Chemotherapy-Erlotinib
Number analyzed (Participants) | 21 | 24
participants
  With any adverse events (AEs) | 14 | 12
  With any serious AEs (SAEs) | 0 | 1
  With any AEs Grade ≥ 3 | 5 | 2
  With any drug related (possible/probable) AEs | 10 | 9
  With any drug related (possible/probable) SAEs | 0 | 0
  With any AEs leading to study drug withdrawal | 0 | 0
  With any AEs leading to death | 0 | 0
  With AEs of Special Interest | 0 | 0
  With pregnancy | 0 | 0

ADVERSE EVENTS:
Time Frame: start of second-line treatment to data cut-off in December 2014 (within 12 months)
Arm/Group | Erlotinib-Chemotherapy | Chemotherapy-Erlotinib
Serious Adverse Events (participants affected / at risk) | 0/21 | 1/24
Other Adverse Events (participants affected / at risk) | 14/21 | 12/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erlotinib-Chemotherapy (N=21) | Chemotherapy-Erlotinib (N=24)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erlotinib-Chemotherapy (N=21) | Chemotherapy-Erlotinib (N=24)
Nausea (Gastrointestinal disorders) | 6 (9) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 4 (14)
Vomiting (Gastrointestinal disorders) | 3 (6) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 8 (8)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Leukopenia (Blood and lymphatic system disorders) | 4 (6) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3 (6) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (4) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (4) | 1 (1)
Platelet count decreased (Investigations) | 2 (3) | 1 (1)
White blood cell count decreased (Investigations) | 3 (6) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (5) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.